CLINICAL TRIAL: NCT01707199
Title: Efficacy and Safety of Artesunate+Sulphadoxine-Pyrimethamine for the Treatment of Uncomplicated Plasmodium Falciparum Malaria in Malaria Control Center Asadabad in Kunar Province of Afghanistan
Brief Title: SPK Study in Afghanistan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: World Health Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPK
Record Dates: First submitted 2012-10-11; First posted 2012-10-16 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Uncomplicated P. Falciparum Malaria
Keywords: P. falciparum; Sulphadoxine-pyrimethamine; Artesunate; Artemisinin Combination Therapy (ACT)
MeSH Terms: interventions — Artesunate; fanasil, pyrimethamine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Artesunate + Sulphadoxine-pyrimethamine (Experimental): AS+SP will be administered according to the patient's age, based on a dose of 4mg artesunate/kg body weight once daily for 3 days plus SP at a dose of 25mg sulphadoxine/kg body weight single dose on the first day.
  One co-blister pack of Artecospe will be used per patient and obtained via WHO from Guilin Pharmaceutical Co. Ltd., Shanghai China, with appropriate expiry date.
  Interventions: Drug: Artesunate + Sulphadoxine-pyrimethamine

INTERVENTIONS:
Drug: Artesunate + Sulphadoxine-pyrimethamine — AS+SP will be administered according to the patient's age, based on a dose of 4mg artesunate/kg body weight once daily for 3 days plus SP at a dose of 25mg sulphadoxine/kg body weight single dose on the first day.
  One co-blister pack of Artecospe will be used per patient and obtained via WHO from Guilin Pharmaceutical Co. Ltd., Shanghai China, with appropriate expiry date.

SUMMARY:
In Afghanistan, studies over the past 15 years have shown a high degree of Plasmodium falciparum resistance to chloroquine. In 2003 the high failure rate of chloroquine against falciparum malaria led the national malaria treatment programme to switch its recommended first line drug treatment for uncomplicated Plasmodium falciparum malaria to artemisinin-based combination therapy (ACT) in the form of Artesunate/Sulphadoxine-Pyrimethamine (AS+SP). Second line drug treatment is oral quinine (7 days).

For operational reasons, prior to recent studies (manuscript in preparation) there have been no molecular data on P. falciparum SP resistance markers from within the borders of Afghanistan. These studies have revealed early evidence of increasing SP resistance (resistance polymorphisms with double DHFR & triple DHPS mutations). The aim of this study is to conduct a focused, prospective study in Kunar for monitoring of the efficacy of the AS+SP combination in this province, along with molecular studies of isolates from recruited patients.

DETAILED DESCRIPTION:
Afghanistan is a poor country that remains largely dependent on foreign aid. Life expectancy remains in the order of 60 years, with 30% of mortality due to communicable diseases.

Malaria is a large health burden, and antimalarial drug resistance poses a considerable threat to malaria control. Resistance to chloroquine was evident in Afghanistan by the late-1990s, with failure rates more than 60% for the country as a whole and as high as 90% for Jalalabad (Nangarhar province). The combination of artesunate with amodiaquine also proved to have low efficacy. In 2004 failure rates for SP for the treatment of P. falciparum were 10-15% consistent with comparable clinical data in Afghan refugees residing in Pakistan. Given this efficacy, the Ministry of Public Health, in consultation with WHO and other international partners, has implemented AS+SP as first-line treatment of slide confirmed P. falciparum malaria in Afghanistan. Quinine (7 days po) is second line treatment. CQ+SP has been the recommended treatment for patients with a presumptive diagnosis of malaria since 2003. Both artesunate and sulphadoxine-pyrimethamine are safe and well tolerated drugs and there is no evidence of an interaction between them.

Artesunate (AS) has been reported to be associated with mild gastrointestinal disturbances, dizziness and tinnitus although none of these associations are convincing. The only potentially serious adverse effect that has been reported with the artemisinin class of drugs in clinical trials is type I hypersensitivity reactions (about 1:3,000 patients). Transient reticulocytopenia, neutropenia, and elevated liver enzyme values have been reported but none have been clinically significant. The weight of evidence suggests these drugs have no significant adverse cardiovascular effects. A variety of clinical, neurophysiological, and pathologic studies in humans have not shown evidence of neurological toxicity. Because these drugs have not been evaluated extensively in early pregnancy in humans, they should be avoided in patients in the first trimester of pregnancy with uncomplicated malaria until more information is available (WHO guidelines 2006).

Sulphadoxine-pyrimethamine (SP) is a fixed combination of a long-acting sulfonamide and the antifolate pyrimethamine. These are synergistic against sensitive parasites. Minor adverse effects are unusual and serious sulfonamide toxicity is very unusual with a single-dose treatment of malaria. The anti-folate properties of pyrimethamine rarely produce toxicity.

The combination of AS + SP has been evaluated extensively in adults and children with uncomplicated malaria and is sufficiently efficacious in areas where 28-day cure rates with sulphadoxine-pyrimethamine alone exceed 80%. This ACT is currently being used in parts of South America, the Middle East, and South Asia where SP susceptibility remains high. Studies conducted between 2004-2006 to evaluate the efficacy of artesunate plus sulphadoxine-pyrimethamine (AS+SP) against P. falciparum showed high efficacy in terms of adequate clinical and parasitological response (Afghanistan National Malaria Strategic Plan).

The genetic determinants of in vitro resistance to the two drug components of SP individually are shown to be point mutations at seven sites in the dihydrofolate reductase gene (dhfr) causing resistance to pyrimethamine and five sites in the dihydropteroate synthase (dhps) gene causing resistance to sulphadoxine. Different combinations of mutations within each gene confer differing degrees of insensitivity. Due to administrative instability, until recently few molecular data relating to P. falciparum SP resistance markers have been available from within the borders of Afghanistan. However the investigators have obtained recent (submitted) data showing that in addition to two resistance polymorphisms in DHFR (C59R and S108N) that are well known to be at high frequency in the region, a small number of parasites in the Kunar province have three mutations (A437G, K540E and A581G) in DHPS.

This study is a prospective, open label, single arm clinical trial to test the PCR confirmed efficacy and tolerability of AS+SP for the treatment of uncomplicated falciparum malaria in Afghanistan. Follow-up will be for 42 days, in order to sensitively detect recrudescence. Recrudescence will be distinguished from re-infection by molecular techniques based on well characterized microsatellite markers msp1, msp2 and glurp will be used. Baseline and any recurrent parasites will be tested for DHFR and DHPS polymorphisms by RFLP as well as sequencing if indicated. The proposed study will provide accurate data and accurate evidences on efficacy of the current malaria treatment regimen in Afghanistan.

ELIGIBILITY:
Inclusion Criteria:

* Males: age over 4 months;
* Females: age 4 months - 11 years inclusive, or 18 years or older;
* Infection with P. falciparum detected by microscopy at a level of 500-150,000/µL asexual forms;
* Presence of axillary or tympanic temperature ≥ 37.5 °C or oral or rectal temperature of ≥ 38 °C or history of fever during the past 24 h;
* ability to swallow oral medication;
* ability and willingness to comply with the study protocol for the duration of the study and to comply with the study visit schedule; and
* Informed consent from the patient or from a parent or guardian in the case of children under 16 years of age.

Exclusion Criteria:

* Presence of general danger signs in children aged under 5 years or signs of severe falciparum malaria according to the definitions of WHO (Appendix 1);
* Infection with another Plasmodium species detected by microscopy not mixed with falciparum;
* Females 18 years or older: a positive pregnancy test or absence of a negative pregnancy test when a pregnancy test is not possible for cultural reasons;
* Breastfeeding
* Presence of severe malnutrition (defined as a child whose growth standard is below -3 z-score, has symmetrical oedema involving at least the feet or has a mid-upper arm circumference < 110 mm);
* Presence of febrile conditions due to diseases other than malaria (e.g. measles, acute lower respiratory tract infection, severe diarrhoea with dehydration) or other known underlying chronic or severe diseases (e.g. cardiac, renal and hepatic diseases, HIV/AIDS);
* Regular medication, which may interfere with antimalarial pharmacokinetics;
* History of hypersensitivity reactions or contraindications to any of the study medications;

Min Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Adequate clinical and parasitological response (ACPR) | 42 days
  WHO defined ACPR

SECONDARY OUTCOMES:
Adverse events | 42 days
  The incidence of any adverse event will be documented. All patients will be asked routinely about previous symptoms and about symptoms that have emerged since the previous follow-up visit.
Molecular markers for antimalarial drug resistance | Baseline
  To study polymorphisms in PfDHFR, PfDHPS and copy number of PfGCH1 which are considered as markers of resistance to Sulphadoxine-pyrimethamine (SP) components.

CONTACTS AND LOCATIONS:
Overall Officials: Ghulam Rahim Awab, MD, Principal Investigator — Research Dept. Ministry of Public Health (MoPH) Afghanistan
Locations (1):
- Narang, Asadabad, Watapoor district health centres, Khāş Kunaṟ, Kunar, Afghanistan

REFERENCES:
- [Derived] Awab GR, Imwong M, Pukrittayakamee S, Alim F, Hanpithakpong W, Tarning J, Dondorp AM, Day NP, White NJ, Woodrow CJ. Clinical trials of artesunate plus sulfadoxine-pyrimethamine for Plasmodium falciparum malaria in Afghanistan: maintained efficacy a decade after introduction. Malar J. 2016 Feb 25;15:121. doi: 10.1186/s12936-016-1167-z. PMID 26917051